CLINICAL TRIAL: NCT02076334
Title: Effect of Compression Garments on Exercise Performance Following Acute High Intensity Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Rhodia, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 13-3101
Record Dates: First submitted 2014-02-24; First posted 2014-03-03 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-04

CONDITIONS: Muscle Damage
Keywords: compression, isokinetic, far-infrared
MeSH Terms: interventions — Polyurethanes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Compression + normal garment (Active Comparator): Far Infrared Fabric during exercise + Spandex at night
  Interventions: Other: Far Infrared Fabric; Other: Spandex
- Normal Garment + Test garment at night (Active Comparator): Spandex during exercise + Far Infrared Fabric at night
  Interventions: Other: Far Infrared Fabric; Other: Spandex
- Normal Garment + normal garment (Sham Comparator): Spandex during exercise + Spandex at night
  Interventions: Other: Spandex
- Test garment + Test garment (Active Comparator): Far Infrared Fabric during exercise + Far Infrared Fabric at night
  Interventions: Other: Far Infrared Fabric

INTERVENTIONS:
Other: Far Infrared Fabric
  Arms: Compression + normal garment; Normal Garment + Test garment at night; Test garment + Test garment
Other: Spandex
  Arms: Compression + normal garment; Normal Garment + Test garment at night; Normal Garment + normal garment

SUMMARY:
To examine the influence of compression garments manufactured with Far-Infrared technology on exercise performance during and after repeated eccentric isokinetic muscle actions of the leg extensors.

DETAILED DESCRIPTION:
Participants: Eighty recreationally active (1-5 hrs per week) healthy participants between the ages of 18 - 35 will visit the Neuromuscular Research Laboratory on 6 separate occasions, with 4 of those occasions also requiring a visit to Health services for a blood draw.

Procedures (methods): During pre-screening, each participant will complete an informed consent document, a health history questionnaire, and have their stature and body mass assessed. A familiarization session will then be conducted on a separate day where all participants will practice the strength assessment, eccentric isokinetic protocol, and ultrasound assessments. Participants will be assigned to 1 of the 4 treatment groups based on their initial maximal isometric strength values using a matched-participants design. The first experimental session will then begin 2-10 days later, where the participants will perform the repeated eccentric exercise protocol (10 sets of 15 eccentric contractions 210 deg/sec with 3 min of rest between sets) with the non-dominant leg following a 60 min rest period where they will wear the apparel and perform a 5 min warm-up on a cycle ergometer. Follow-up blood draws and strength and ultrasound assessments will be obtained at 24 and 48 hours post-exercise. Each participant will also complete a visual analog scale at baseline, 24, 48, and 72 hours post-exercise to examine perceived muscle soreness.

ELIGIBILITY:
Inclusion Criteria:

* Cohort of Adult Males & Females
* Participant is between the ages of 18-35
* Healthy, Recreationally Active (1-5 hours per week)
* Participant has provided written and dated informed consent to participate in the study
* Participant is apparently healthy and free from disease, as determined by a health history questionnaire
* Participant agrees to abstain from smoking, caffeine (4hrs prior), tobacco (24hrs prior), and alcohol (24 hrs) before testing days
* Participant agrees to abstain from exercise 24 hours prior to each testing visit and after 72 hours of the induced exercise damage
* Participant will refrain from the use of non-steroidal anti-inflammatory drugs (NSAIDs) and protein supplementation 24 hours before the exercise testing protocol, as well as for the 72 hour period following the exercise testing protocol.

Exclusion Criteria:

* Participant is using, or has used one of the following dietary supplements within 12 weeks prior to enrollment: beta-alanine, creatine, taurine, or any supplemental antioxidants (Acai, pomegranate, beet juice).
* Participant is in, or has participated in another clinical trial within 6 weeks prior to enrollment
* Participant has a known allergy or sensitivity to test product (determined from health history questionnaire and consent form)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbie Smith-Ryan, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Exercise and Sport Science (University of North Carolina), Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/19222900

RESULTS

PARTICIPANT FLOW:
Groups:
- Compression + Normal Garment: Far Infrared Fabric during exercise + Spandex at night
  Far Infrared Fabric
  Spandex
- Normal Garment + Test Garment at Night: Spandex during exercise + Far Infrared Fabric at night
  Far Infrared Fabric
  Spandex
- Normal Garment + Normal Garment: Spandex during exercise + Spandex at night
  Spandex
- Test Garment + Test Garment: Far Infrared Fabric during exercise + Far Infrared Fabric at night
  Far Infrared Fabric
Period: Overall Study
Arm/Group | Compression + Normal Garment | Normal Garment + Test Garment at Night | Normal Garment + Normal Garment | Test Garment + Test Garment
Started | 21 | 21 | 21 | 21
Completed | 20 | 20 | 20 | 20
Not Completed | 1 | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — muscle soreness | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compression + Normal Garment | Normal Garment + Test Garment at Night | Normal Garment + Normal Garment | Test Garment + Test Garment | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 20 | 80
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 20.5 (1.4) | 20.9 (2.0) | 22.1 (3.2) | 21.0 (2.5) | 21 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 12 | 12 | 50
  Male | 8 | 6 | 8 | 8 | 30
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80

OUTCOME MEASURES:

1. Primary Outcome: Maximal Voluntary Contraction (MVC)
Time Frame: up to 72 hours
Measure: Mean (Standard Deviation); unit: Newton-meters
Arm/Group | Compression + Normal Garment | Normal Garment + Test Garment at Night | Normal Garment + Normal Garment | Test Garment + Test Garment
Number analyzed (Participants) | 20 | 20 | 20 | 20
Newton-meters | 182.4 (45.7) | 198.7 (56.2) | 208 (70.5) | 186.4 (44.1)

2. Secondary Outcome: Creatine Kinase
Time Frame: baseline, 24 hrs and 48 hrs post
Measure: Mean (Standard Error); unit: u/L
Arm/Group | Compression + Normal Garment | Normal Garment + Test Garment at Night | Normal Garment + Normal Garment | Test Garment + Test Garment
Number analyzed (Participants) | 20 | 20 | 20 | 20
u/L
  Baseline | 140.6 (40.4) | 158.2 (41.5) | 181.2 (40.4) | 108.2 (41.5)
  24 H post | 277.1 (102.6) | 458.5 (105.2) | 516.2 (102.6) | 332.8 (105.2)
  48 H post | 225.8 (127.3) | 355.8 (130.6) | 542.9 (127.3) | 263.6 (130.6)

ADVERSE EVENTS:
Time Frame: Duration of study enrollment (3 weeks)
Arm/Group | Compression + Normal Garment | Normal Garment + Test Garment at Night | Normal Garment + Normal Garment | Test Garment + Test Garment
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No